CLINICAL TRIAL: NCT06022302
Title: Effects of Changing Intestinal Transit Time on Gut Microbial Composition and Metabolism During a Dietary Intervention with Low and High Fiber.
Brief Title: Effects of Changing Intestinal Transit Time on Gut Microbial Composition and Metabolism
Acronym: PRIMA-KOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Technical University of Denmark (Other); KU Leuven (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Henrik Munch Roager, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M245
Record Dates: First submitted 2023-08-11; First posted 2023-09-01 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Diet, Healthy; Metabolic Disease
Keywords: Microbiome; Metabolomics; Transit time; Nutrition; Dietary fibre
MeSH Terms: conditions — Metabolic Diseases | interventions — Diet; Laxatives

STUDY DESIGN:
Intervention Model Description: Overall, there are two parallel arms (low- and high-fiber diet) to which the participants will be randomized with an allocation ratio 1:1. In each arm participants will be exposed to a crossover design where participants in random order will continue on the meal intervention alone (control) or receive Movicol (a laxative) along with the meal intervention to shorten intestinal transit time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-fiber diet (Experimental): The high-fiber diet will consist of foods rich in dietary fiber such as coarse vegetables, wholegrain bread, and fruits representing a broad range of dietary fibers aiming for ≈40 g of fiber/10 MJ.
  Interventions: Drug: Diet + laxative; Other: Diet only
- Low-fiber diet (Experimental): The low-fiber diet will consist of foods poor in fiber such as white bread and refined foods aiming for ≈10 g of fiber/10 MJ.
  Interventions: Drug: Diet + laxative; Other: Diet only

INTERVENTIONS:
Drug: Diet + laxative — The participants will start by consuming one sacket of Movicol powder (13 g macrogol 3350) on the first day. On day 2, the participants will consume two sackets of Movicol powder (26 g macrogol 3350), one with breakfast in the morning and one before sleep in the evening. The participants will continue consuming two sackets per day (one morning, one evening) until the following study visit, day 8 (seven days in total). If the participants have a very loose stomach (recorded as Bristol stool scale ≥6), they will be instructed to reduce Movicol by one sacket/day. In case the participants have not passed a stool on day 2 or in the morning of day 3, the participants will increase the dose to a maximum of three sackets of Movicol powder (39 g macrogol 3350) per day (morning, noon, and evening) and continue this until the following study visit at day 8. If three sackets cause very loose stomach the participants will decrease the number of sackets consumed.
Other: Diet only — This is only a control and participants will not receive Movicol.
  Other Names: Control

SUMMARY:
The aim of this study is to investigate how a short versus a long transit time impacts the gut microbiome's response to a high-fiber and a low-fiber diet, respectively. Such insights could help us understand personal responses to diets and be a first step towards personalized dietary recommendations targeting the gut microbiome.

DETAILED DESCRIPTION:
The study consists of two parallel arms of whole-meal diets, a low-fiber diet, and a high-fiber diet, respectively. Each arm is designed as a cross-over where participants, in random order, are administered a laxative (Movicol) along with the provided diet to shorten their intestinal transit time or simply consume the provided whole-meal diet (control).

The two intervention periods both involve the following:

* One week of run-in where participants consume the provided whole-meal diet.
* One week where participants either consume Movicol with the provided whole-meal diet or simply continue consuming the provided whole-meal diet (control).

Both arms begin with a screening visit and one week where participants consume and record their habitual diets. Subsequently, the first intervention period follows with one visit before and after each of the two weeks (visit 1-3) followed by the second intervention period with one visit before and after each of the two weeks (visit 4-6). The two cross-over periods are split by a washout of at least two weeks.

The study thus runs for approximately 7-8 weeks depending on the length of the washout and consists of seven visits (one screening visit and six regular visits) in total.

ELIGIBILITY:
Inclusion Criteria:

* 18.5-30.0 kg/m2 BMI
* Self-reported ≤3.5 spontaneous bowel movements per week
* Willing to collect urine and stool samples at home and able to temporarily store them in their own freezer in a provided container.
* Willing to eat the foods provided.
* Owns a smartphone (iOS 11.0 and later or Android 5.0 and up) with access to the internet.

Exclusion Criteria:

* Pregnant or lactating women.
* Diagnosis of irritable bowel syndrome (IBS), small intestinal bacterial overgrowth (SIBO), inflammatory bowel diseases (IBD), Gastrointestinal obstruction, or Ischemic colitis
* Diagnosed constipation according to the ROME IV criteria
* Intake of antibiotics ˂ 1month, or any medication that can affect the outcomes of the study
* Regular use of diarrhea inhibitors or laxatives
* Dysphagia
* Any chronic disease that can affect the outcomes of the study or pose a risk when consuming Movicol
* Intake of medications potentially altering gastric pH (proton pump inhibitors, histamine receptor antagonists, antacids)
* Intake of medications potentially altering the gastrointestinal motility (prokinetics, antiemetic agents, anti-cholinergic agents, narcotic analgetics, nonsteroidal anti-inflammatory drugs, and peroral glucocorticoids)
* Concurrent participation in another trial
* Any condition that makes the project responsible researcher to doubt the feasibility of the volunteer´s participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Fecal butyrate over urine p-cresol sulfate ratio | From visit 1 through to study completion, an average of 7 weeks
  Changes in ratio between fecal butyrate (reflecting saccharolytic fermentation) and urine p-cresol sulfate (reflecting proteolytic fermentation) between interventions.

SECONDARY OUTCOMES:
Whole gut transit time measured by sweet corn | From visit 1 through to study completion, an average of 7 weeks
  Changes in whole gut transit time between interventions determined by the passage time of sweet corn.
Whole gut transit time measured by blue muffins | From visit 1 through to study completion, an average of 7 weeks
  Changes in whole gut transit time between interventions determined by the passage time of muffins with blue dye.
Stool consistency | From visit 1 through to study completion, an average of 7 weeks
  Changes in stool consistency determined by Bristol Stool Scale. The Bristol Stool Scale measures stool consistency on a scale from 1-7 with high numbers reflecting loose stool.
Change in bowel movement frequency | From visit 1 through to study completion, an average of 7 weeks
  Changes in bowel movement frequency will be measured by the participants recording every bowel movement in a defecation diary during the study.
Fecal water content in percentage of stool weight | From visit 1 through to study completion, an average of 7 weeks
  Change in fecal water content between interventions.
Fecal concentration of short-chain fatty acids | From visit 1 through to study completion, an average of 7 weeks
  Change in concentration of short-chain fatty acids between interventions.
Fecal pH | From visit 1 through to study completion, an average of 7 weeks
  Change in fecal pH level between interventions.
Fecal ammonia concentration | From visit 1 through to study completion, an average of 7 weeks
  Change in ammonia content between interventions.
Concentration of fasting plasma short-chain fatty acids | From visit 1 through to study completion, an average of 7 weeks
  Change in concentration of short-chain fatty acids between interventions.
Fasting plasma concentrations of bile acids | From visit 1 through to study completion, an average of 7 weeks
  Change in concentration of bile acids in fasting blood between interventions.
Fasting breath methane and hydrogen levels in parts per million | From visit 1 through to study completion, an average of 7 weeks
  Changes in fasting breath methane and hydrogen concentration measured in parts per million (PPM) in exhalations between interventions.
Microbial metabolites in urine from proteolytic fermentation as assessed by mass spectrometry | From visit 1 through to study completion, an average of 7 weeks
  Changes in the urine concentration of metabolites of microbial proteolysis between interventions.
Microbial metabolites in blood from proteolytic fermentation as assessed by mass spectrometry | From visit 1 through to study completion, an average of 7 weeks
  Changes in the blood concentration of metabolites of microbial proteolysis between interventions.
Fecal metabolome as assessed by untargeted metabolomics | From visit 1 through to study completion, an average of 7 weeks
  Changes in the fecal metabolome between interventions.
Gut microbiome assessed by shotgun sequencing | From visit 1 through to study completion, an average of 7 weeks
  Changes in gut microbiota composition between interventions.
Gut microbiome assessed by 16S amplicon sequencing | From visit 1 through to study completion, an average of 7 weeks
  Changes in gut microbiota composition between interventions.

OTHER OUTCOMES:
Urine metabolome as assessed by untargeted metabolomics | From visit 1 through to study completion, an average of 7 weeks
  Changes in the urine metabolome between interventions.
Blood metabolome as assessed by untargeted metabolomics | From visit 1 through to study completion, an average of 7 weeks
  Changes in the blood metabolome between interventions.
Fecal microbial metabolites of proteolytic fermentation measured by mass spectrometry | From visit 1 through to study completion, an average of 7 weeks
  Assessment of changes in fecal microbial metabolites of proteolytic fermentation (amino acid-derived metabolites).
Fecal enzymatic activities | From visit 1 through to study completion, an average of 7 weeks
  Assessment of changes in enzymatic activities measured in fecal samples between interventions.
Fecal residual carbohydrate concentration | From visit 1 through to study completion, an average of 7 weeks
  Change in residual carbohydrate concentration measured in fecal samples between interventions.
Fecal energy density | From visit 1 through to study completion, an average of 7 weeks
  Change in fecal energy density measured by bomb calorimetry in fecal samples between interventions.
Fecal redox potential measured in mV | From visit 1 through to study completion, an average of 7 weeks
  Change in redox potential measured in fecal samples between interventions.
Fecal carbon:nitrogen (C:N) ratio | From visit 1 through to study completion, an average of 7 weeks
  Change in C:N ratio measured in fecal samples between interventions.
Fecal microbial load (cells per gram) | From visit 1 through to study completion, an average of 7 weeks
  Change in microbial load in fecal samples between interventions.
Fecal calprotectin concentration | From visit 1 through to study completion, an average of 7 weeks
  Change in concentration of calprotectin measured in fecal samples between interventions. Used as a measure of intestinal inflammation.
Change in various markers related to glucose metabolism | From visit 1 through to study completion, an average of 7 weeks
  Changes in the concentration of various standard markers of glucose metabolism in fasting blood samples between interventions.
Change in various markers related to lipid metabolism | From visit 1 through to study completion, an average of 7 weeks
  Changes in concentration of various standard biochemical markers of lipid metabolism in fasting blood samples between interventions.
Change in various markers of inflammation | From visit 1 through to study completion, an average of 7 weeks
  Change in concentration of various inflammatory markers in fasting blood between interventions.
Change in various appetite hormones | From visit 1 through to study completion, an average of 7 weeks
  Change in concentration of various appetite hormones in fasting blood between interventions.
Urinary creatinine concentration | From visit 1 through to study completion, an average of 7 weeks
  Measurement of urinary levels of creatinine from spot urine samples between interventions.
Amylase gene copy number | At visit 1
  Measurement of amylase gene copy numbers from blood samples at visit 1 to determine the phenotype of the participants.
Change in body weight | From baseline through to study completion, an average of 8 weeks
  Change in body weight is measured using a calibrated digital scale to ensure/monitor weight stability throughout the study.
Measurement of breath hydrogen and methane profiles in parts per million (Area under the curve) | From baseline through to study completion, an average of 8 weeks
  Measurement of the hydrogen and methane concentrations, in parts per million (PPM), in morning, noon, and evening breath exhalations every day during the study using a portable breath analyzer.
Habitual dietary intake | Before each intervention, 6 days in total
  Habitual dietary intake will be measured two times over 3 days each using an online 24h dietary record MyFood24 prior to visit 1 and 4.
Change in self-perceived stress level | At visit 1 and after each intervention
  Participants' stress levels will be assessed using Cohen's 10-item Perceived Stress Scale (PSS) at visits 1, 3, and 6. Each item is scored on a scale from 1-5 where higher values represent a higher level of self-perceived stress.
Change in subjective gastrointestinal symptoms | From visit 1 through to study completion, an average of 7 weeks
  Changes in subjective gastrointestinal symptoms reported by participants on a visual analog scale from 0 to 10, where 0 means no symptoms and 10 means the worst possible symptoms. The questionnaire includes the following symptoms: overall stomach and intestinal symptoms, stomachache, flatulence, bloating, constipation, and diarrhea.
Physical activity level | At baseline
  Physical activity will be measured by the International Physical Activity Questionnaire short form (IPAQ-s) at the screening visit. The IPAQ-s consists of 7 items asking about the amount of physical activity (in minutes) at different intensities. The score is the sum of minutes of activity at each intensity level given as metabolic equivalents (METs). The higher the MET score, the more physically active the participant is.
Change in sleep quality | At visit 1 and after each intervention
  Changes in sleep pattern and quality will be measured by the Pittsburg Sleep Quality Index (PSQI) at visits 1, 3, and 6. The PSQI consists of 19 items, summed into seven component scores and one overall composite score. Each item is rated on a scale from 0-3 with lower scores reflecting healthier sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Department of Nutrition, Exercise and Sports, Copenhagen, Denmark